CLINICAL TRIAL: NCT02914587
Title: Computer-Assisted Hair Implantation Using ARTAS System VS Manual Implantation Technique Hair Restoration Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Restoration Robotics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CP-003
Record Dates: First submitted 2016-09-19; First posted 2016-09-26 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Androgenic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARTAS System (Experimental): Implantation with the ARTAS System.
  Interventions: Device: ARTAS System
- Manual Implantation (Active Comparator): Implantation manually.
  Interventions: Other: Manual Implantation

INTERVENTIONS:
Device: ARTAS System
  Arms: ARTAS System
Other: Manual Implantation
  Arms: Manual Implantation

SUMMARY:
To investigate and compare the safety and effectiveness of the ARTAS™ System to manual hair follicle implantation method following a nine month period of post-procedure evaluation.

DETAILED DESCRIPTION:
This comparative study is a multi-center, prospective, blinded, randomized controlled clinical study where subjects act as their own control.

The purpose of this study is to demonstrate that the ARTAS System is safe and effective for implanting follicular hair units.

Patients will be followed for a nine months period of time.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male with clinical diagnosis of androgenetic alopecia with Norwood-Hamilton grade of IV-VI;
* Subject is 29 to 70 years old;
* Subject has black or brown hair color;
* Subject has straight hair;
* Subject agrees to cut hair short (about 1-1.4 mm) on the scalp in the designated study areas for harvesting and implantation;
* Subject agrees to have 6 dot tattoos placed on scalp;
* Subject is able to understand and provide written consent; and
* Subject consents to post-operative follow-up per protocol.

Exclusion Criteria:

* Subject has prior history of scalp reduction surgery(s);
* Subject has prior history of hair restoration procedure(s) using the strip excision technique;
* Subject has bleeding diathesis;
* Subject has active use of anti-coagulation medication;
* Subject has used finasteride in the previous 6 months, or plans to use finasteride during the study;
* Subject has used minoxidil in the previous 2 weeks, or plans to use minoxidil during the study; or
* Subject has any other condition that, in the opinion of the investigator, makes the subject inappropriate to take part in this study.

Ages: 29 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08; Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Hair Survival rate 9-months post procedure | 9 month
  Hair survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Berman Skin Institute, Palo Alto, California, United States